CLINICAL TRIAL: NCT01925937
Title: Atorvastatin/CoenzymeQ10 in Congestive Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amin Nemati, member of Isfahan Medical Students Research Committee, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 392219
Record Dates: First submitted 2013-08-08; First posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Congestive Heart Failure
Keywords: Coenzyme Q10; Atorvastatin; clinical trial; congestive heart failure
MeSH Terms: conditions — Heart Failure | interventions — Atorvastatin; coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Coenzyme Q10 & Atorvastatin (Experimental): 10 mg Atorvastatin daily plus 100 mg Coenzyme Q10 pearl supplement twice daily for four months.
  Interventions: Drug: Atorvastatin; Drug: Coenzyme Q10
- Atorvastatin & placebo (Active Comparator): 10 mg Atorvastatin daily and the placebo of Coenzyme Q10 pearl for four months.
  Interventions: Drug: Atorvastatin; Drug: placebo for coenzyme Q10

INTERVENTIONS:
Drug: Atorvastatin
Drug: Coenzyme Q10
  Arms: Coenzyme Q10 & Atorvastatin
Drug: placebo for coenzyme Q10
  Arms: Atorvastatin & placebo

SUMMARY:
The aim of this study is to compare the effect of addition of combination of Atorvastatin/CoenzymeQ10 to standard congestive heart failure (CHF) treatment versus addition of Atorvastatin alone on CHF outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Documented Congestive hear failure
* Ejection Fraction less than 40 percent
* Compensated heart failure without hospital admission during previous three months
* No change in type and dose of medications in the last months
* New York Heart Association Function Class 2 to 4

Exclusion Criteria:

* Acute coronary syndrome developing in the last month
* Active myocarditis
* Active pericarditis
* Uncontrolled hypertension
* Hepatic failure(Child B,C)
* Pulmonary failure
* Renal failure
* Heart failure with KILLIP classification 3 and 4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac Ejection Fraction (EF) | Baseline for the first time and after 4 months for the second time
  For the determination of change in EF,cardiac EF was determined two times . Baseline :at the beginning of study(before intervention) and the second time after 4 months(after intervention).

SECONDARY OUTCOMES:
Change in New York Heart Association Function Class | Baseline for the first time and after 4 months for the second time
  For the determination of change in New York Heart Association Function Class.it was determined two times .Baseline:at the beginning of study(before intervention)and the second time after 4 months(after intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Pourmoghaddas, cardiologist, Study Director — Isfahan Cardiovascular Research Institute, Isfahan University of Medical Sciences, Isfahan, Iran.
Locations (1):
- Vice Chancellery for Research of Isfahan University of Medical Sciences, Isfahan, Iran, Isfahan, Isfahan, Iran